CLINICAL TRIAL: NCT06816173
Title: Effect of Propofol Versus Remimazolam Intravenous Anesthesia Combined With Regional or Caudal Block on Respiratory Depression in Young Children: A Randomized Controlled Clinical Study
Brief Title: Effect of Propofol Versus Remimazolam Intravenous Anesthesia on Respiratory Depression
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Second Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SAHoWMU-CR2025-03-102
Record Dates: First submitted 2025-02-04; First posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Respiratory Depression
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group P（Propofol group） (Experimental): Patients were assigned to group P (Propofol group) using a computer-generated random number table
  Interventions: Drug: Propofol group
- group R (Remimazolaml group) (Experimental): Patients were assigned to group R (Remimazolaml group) using a computer-generated random number table
  Interventions: Drug: Remimazolam group

INTERVENTIONS:
Drug: Propofol group — Induction phase: Administer fentanyl at a dose of 2-3 mcg/kg, and after 3 minutes, administer propofol intravenously at a dose of 2.0 mg/kg.
  Maintenance phase: Infuse propofol (4-12 mg/kg/h) and maintain a constant infusion of remifentanil at a rate of 0.05-0.4 μg/kg/min. Subsequently, perform regional block (0.25% ropivacaine 0.5 ml/kg) or caudal block (lower limbs or perineal area: 0.25% ropivacaine 0.5 ml/kg; lower abdomen/inguinal area: 0.25% ropivacaine 0.75 ml/kg). After the local anesthetic has taken full effect, stop the infusion of remifentanil.
  Arms: group P（Propofol group）
Drug: Remimazolam group — Induction phase: Administer fentanyl at a dose of 2-3 mcg/kg, and after 3 minutes, administer remimazolam intravenously at a dose of 0.45-0.55 mg/kg.
  Maintenance phase: Infuse remimazolam (1-3 mg/kg/h) and maintain a constant infusion of remifentanil at a rate of 0.05-0.4 μg/kg/min. Subsequently, perform regional block (0.25% ropivacaine 0.5 ml/kg) or caudal block (lower limbs or perineal area: 0.25% ropivacaine 0.5 ml/kg; lower abdomen/inguinal area: 0.25% ropivacaine 0.75 ml/kg). After the local anesthetic has taken full effect, stop the infusion of remifentanil.
  Arms: group R (Remimazolaml group)

SUMMARY:
General anesthesia is the preferred choice for pediatric patients, but the induction of volatile anesthetics via face mask may cause preoperative anxiety and postoperative delirium. Total intravenous anesthesia (TIVA) is more suitable for pediatric patients, as it can effectively alleviate preoperative anxiety, reduce the risk of postoperative delirium and mania, shorten hospital stay, reduce medical burden, and increase parental satisfaction. Propofol, although effective for anesthesia, has drawbacks such as injection pain and respiratory and circulatory suppression. Remimazolam is a novel ultra-short-acting benzodiazepine drug, which has no injection pain, minimal impact on respiration and circulation, and rapid onset and elimination, making it suitable for children. However, research on remimazolam in children is limited. This study aims to compare the effect of propofol and remimazolam intravenous anesthesia combined with regional or caudal block on respiratory depression in preschoolers.

DETAILED DESCRIPTION:
Ninety-six children aged 3-6 years scheduled for surgery under general anesthesia were randomly divided into two groups. Initially, fentanyl was administered at a dose of 2-3 mcg/kg, and after 3 minutes, different test drugs were given according to the group assignment. In group P, propofol was administered intravenously at a dose of 2.0 mg/kg, while in group R, remimazolam was administered intravenously at a dose of 0.45-0.55 mg/kg. After achieving loss of consciousness (LoC, MOAA/S ≤ 1), a laryngeal mask was inserted, and spontaneous breathing was maintained. Subsequently, the test drugs were infused according to the group assignment, and both groups received a constant infusion of remifentanil at a rate of 0.05-0.4 μg/kg/min. After connecting the micro-infusion pump, regional or caudal block was performed. Once the local anesthetic had taken full effect, the infusion of remifentanil was stopped, and surgery began. The test drugs were stopped approximately 5 minutes before the end of the surgery, and the laryngeal mask was removed when spontaneous breathing reached a tidal volume of ≥ 6 ml/kg and a frequency of ≥ 15 breaths per minute.

The following data were recorded: the time to loss of consciousness, the incidence of respiratory depression during anesthesia, the success rate of intravenous sedation, the incidence of postoperative agitation, recovery time, MOAA/S scores, and vital signs such as heart rate, blood pressure, and pulse oximetry.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 3-6 years, gender unrestricted;
2. American Society of Anesthesiologists (ASA) physical status classification of I-II;
3. Body Mass Index (BMI) between 14 kg/m² and 25 kg/m²;
4. Patients requiring elective surgery that can be completely anesthetized through regional or caudal block;
5. The child's parent or legal guardian voluntarily participates in this trial and signs the informed consent form.

Exclusion Criteria:

1. Children requiring special care or under the supervision of a court or social welfare agency;
2. Children who have received general anesthesia within 3 months prior to the screening period;
3. Children with a history of respiratory diseases within the past 2 weeks or those deemed to have difficult airway management: Modified Mallampati score of III or IV;
4. Children with severe cardiovascular diseases or endocrine system abnormalities;
5. Children with known psychiatric disorders or cognitive impairments;
6. Children with abnormal liver function, ALT (alanine aminotransferase) and/or AST (aspartate aminotransferase) >1.5 times the upper limit of normal; children with total bilirubin exceeding the upper limit of normal; children with abnormal kidney function, creatinine and/or blood urea nitrogen higher than the upper limit of normal;
7. Children known or suspected to be allergic to the study drug or benzodiazepines.

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 96 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Incidence of respiratory depression during anesthesia | During the induction and maintenance of anesthesia
  During the induction and maintenance of anesthesia, the occurrence of respiratory depression is defined by meeting at least one of the following criteria:
  1. Spontaneous respiratory rate (RR) less than 12 breaths/min for a duration of 1 minute, or peripheral oxygen saturation (SpO2) less than 92% for a duration of 10 seconds.
  2. Loss of spontaneous breathing.

SECONDARY OUTCOMES:
Success rate of anesthesia induction and maintenance | During the induction and maintenance of anesthesia
  Successful anesthesia induction is defined as achieving loss of consciousness (LoC) without the use of rescue sedation during the induction period. Successful anesthesia maintenance is defined as not requiring rescue sedation or interruption of the study drug during the maintenance period.
Time to Loss of Consciousness (LoC) | During anesthesia induction
  The time from the start of administration of the study drug to the loss of consciousness in the subjects, defined as MOAA/S ≤ 1.
PAED scores of the subjects in the PACU | Assess every 5 minutes after the child regains consciousness.
  The PAED scale consists of 5 items, which are: obeying commands and being communicative, purposeful behavior, attention to the surrounding environment, restlessness, and crying that cannot be comforted. A PAED score of ≥12 is defined as delirium.
Recovery time | The moment of anesthesia recovery
  The time from the cessation of the study drug infusion during anesthesia maintenance to the recovery of the subject (defined as the first time when the MOAA/S score is continuously three times 5).
Time-frequency characteristics of electroencephalogram (EEG) | Intraoperative (during remimazolam general anesthesia (including anesthesia induction, maintenance and recovery)
  The time-frequency characteristics of the frontal electroencephalogram (EEG) in children of different age groups under propofol or remimazolam general anesthesia (including induction, maintenance, and recovery phases).

CONTACTS AND LOCATIONS:
Overall Officials: Huacheng Liu, Principal Investigator — Second Affiliated Hospital of Wenzhou Medical University; Yuhang Cai, Principal Investigator — Second Affiliated Hospital of Wenzhou Medical University
Locations (1):
- The second Affiliated Hospital and Yuying Children's Hospital of Wenzhou Medical University, Wenzhou, Zhejiang, China